CLINICAL TRIAL: NCT01940484
Title: An Observational, Non-Interventional Cohort Study to Observe the Efficacy and Use of MIRCERA in the Treatment of Chronic Renal Anaemia in Patients With Chronic Kidney Disease Stage V on Haemodialysis
Brief Title: An Observational Study of Methoxy Polyethylene Glycol-Epoetin Beta (Mircera) in Stage V Chronic Kidney Disease Participants on Hemodialysis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22344
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Results first posted 2016-04-20 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-05

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Chronic Renal Anemia Participants: Participants with chronic kidney disease and who are on hemodialysis and on methoxy polyethylene glycol epoetin beta as per physician's discretion for treatment of chronic renal anemia will be observed for a period of 6-12 months.
  Interventions: Drug: Methoxy polyethylene glycol epoetin beta

INTERVENTIONS:
Drug: Methoxy polyethylene glycol epoetin beta
  Other Names: Mircera

SUMMARY:
This observational study will evaluate the efficacy and use of Methoxy polyethylene glycol-epoetin beta (Mircera) in participants with Stage V chronic kidney disease on hemodialysis receiving an erythropoietin prior to study entry. Attending physicians should have made the decision of placing the participant on methoxy polyethylene glycol epoetin beta in advance and not related to the study. The therapy will be administered by the attendant treating physician according to specifications in the package insert guidelines and to the routine of the site.

ELIGIBILITY:
Inclusion Criteria:

* Participants with chronic renal anemia with Stage V chronic kidney disease on hemodialysis and with a hemoglobin level of 10.0 - 13.0 grams per deciliter (g/dL)
* Participants had to be receiving an ESA prior to entering the study
* Female participants of childbearing age had to be using effective contraceptive methods

Exclusion Criteria:

* As per approved package insert
* Any contraindication to ESA treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Stage V chronic kidney disease on hemodialysis with renal anemia receiving erythropoiesis-stimulating agent (ESA).
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2009-08-31 (Actual); Primary Completion 2012-07-31 (Actual); Study Completion 2012-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- South Africa (10):
  - Glynnwood Hospital, Benoni
  - Universitas Private Hospital, Bloemfontein
  - GVI Constantiaberg, Cape Town
  - Groote Schuur Hospital; Renal Unit, Cape Town
  - N1City Hospital, Cape Town
  - Dr KB Parag & Raghubir Kidney and Dialysis Centre, Durban
  - St Augustine Hospital / Chelmsford Medical Center; Nephrology, Durban
  - Mayo Clinic, Johannesburg
  - Sunninghill Hospital, Johannesburg
  - Donald Gordon Medical Centre, Johannesburg

RESULTS

PARTICIPANT FLOW:
Groups:
- Chronic Renal Anemia Participants: Participants with chronic kidney disease and who were on hemodialysis and prescribed methoxy polyethylene glycol epoetin beta (Mircera) as per physician's discretion for treatment of chronic renal anemia were observed for a period of 6-12 months.
Period: Overall Study
Arm/Group | Chronic Renal Anemia Participants
Started | 98
Completed | 88
Not Completed | 10
Not completed — Withdrawal by Subject | 3
Not completed — Underwent transplantation | 4
Not completed — Death | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Included all enrolled participants.
Groups:
- Chronic Renal Anemia Participants: Participants with chronic kidney disease and who were on hemodialysis and prescribed methoxy polyethylene glycol epoetin beta as per physician's discretion for treatment of chronic renal anemia were observed for a period of 6-12 months.
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 59
Diastolic blood pressure (DBP) [Mean (Standard Deviation); unit: millimeters of Mercury (mm Hg)] — Participant's baseline DBP is reported before undergoing hemodialysis as 'DBP pre-dialysis' and after undergoing hemodialysis as 'DBP post-dialysis' and "n" represents the number of participants evaluable for the specified baseline measure.
  millimeters of Mercury (mm Hg)
    DBP pre-dialysis (n=95) | 82.5 (13.6)
    DBP post-dialysis (n=93) | 78.8 (13.8)
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mm Hg] — Participant's baseline SBP is reported before undergoing hemodialysis as 'SBP pre-dialysis' and after undergoing hemodialysis as 'SBP post-dialysis' and "n" represents the number of participants evaluable for the specified baseline measure.
  mm Hg
    SBP pre-dialysis (n=95) | 145.7 (18.8)
    SBP post-dialysis (n=93) | 136.7 (19.6)
Pulse rate [Mean (Standard Deviation); unit: beats per minute] — The number of participants analyzed for this baseline measure is 65.
  beats per minute | 73.4 (13.1)
Height [Mean (Standard Deviation); unit: centimeters (cm)] — The number of participants analyzed for this baseline measure is 86.
  centimeters (cm) | 167.5 (10.3)
Body Weight [Mean (Standard Deviation); unit: kilograms] — The number of participants analyzed for this baseline measure is 97.
  kilograms | 75.0 (18.5)
Number of Participants With Hemoglobin Level Within the Range of 11-12 Grams Per Deciliter (g/dL) [Number; unit: participants] | 25
Mean Hemoglobin Value [Mean (Standard Deviation); unit: g/dL] | 11.57 (1.47)
Methoxy Polyethylene Glycol-Epoetin Beta Dose [Mean (Standard Deviation); unit: micrograms (mcg)] — The number of participants analyzed for this baseline measure is 97.
  micrograms (mcg) | 107.47 (41.80)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hemoglobin Values Within the Target Range of 11-12 g/dL at Visit 2 (Month 1)
Time Frame: Visit 2 (Month 1)
Population: Included all enrolled participants who were evaluable for this outcome at the specified timepoint.
Measure: Number; unit: participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 87
participants | 23

2. Primary Outcome: Number of Participants With Hemoglobin Values Within the Target Range of 11-12 g/dL at Visit 3 (Month 2)
Time Frame: Visit 3 (Month 2)
Population: Included all enrolled participants who were evaluable for this outcome at the specified timepoint.
Measure: Number; unit: participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 89
participants | 26

3. Primary Outcome: Number of Participants With Hemoglobin Values Within the Target Range of 11-12 g/dL at Visit 4 (Month 3)
Time Frame: Visit 4 (Month 3)
Population: Included all enrolled participants who were evaluable for this outcome at the specified timepoint.
Measure: Number; unit: participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 86
participants | 22

4. Primary Outcome: Number of Participants With Hemoglobin Values Within the Target Range of 11-12 g/dL at Visit 5 (Month 4)
Time Frame: Visit 5 (Month 4)
Population: Included all enrolled participants who were evaluable for this outcome at the specified timepoint.
Measure: Number; unit: participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 83
participants | 17

5. Primary Outcome: Number of Participants With Hemoglobin Values Within the Target Range of 11-12 g/dL at Visit 6 (Month 5)
Time Frame: Visit 6 (Month 5)
Population: Included all enrolled participants who were evaluable for this outcome at the specified timepoint.
Measure: Number; unit: participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 86
participants | 24

6. Primary Outcome: Number of Participants With Hemoglobin Values Within the Target Range of 11-12 g/dL at Visit 7 (Month 6)
Time Frame: Visit 7 (Month 6)
Population: Included all enrolled participants who were evaluable for this outcome at the specified timepoint.
Measure: Number; unit: participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 78
participants | 24

7. Primary Outcome: Mean Hemoglobin Value at Visit 2 (Month 1)
Time Frame: Visit 2 (Month 1)
Population: Included all enrolled participants who were evaluable for this outcome at the specified timepoint.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 87
g/dL | 11.31 (1.74)

8. Primary Outcome: Mean Hemoglobin Value at Visit 3 (Month 2)
Time Frame: Visit 3 (Month 2)
Population: Included all enrolled participants who were evaluable for this outcome at the specified timepoint.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 89
g/dL | 10.81 (1.75)

9. Primary Outcome: Mean Hemoglobin Value at Visit 4 (Month 3)
Time Frame: Visit 4 (Month 3)
Population: Included all enrolled participants who were evaluable for this outcome at the specified timepoint.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 86
g/dL | 10.61 (1.63)

10. Primary Outcome: Mean Hemoglobin Value at Visit 5 (Month 4)
Time Frame: Visit 5 (Month 4)
Population: Included all enrolled participants who were evaluable for this outcome at the specified timepoint.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 83
g/dL | 10.80 (1.77)

11. Primary Outcome: Mean Hemoglobin Value at Visit 6 (Month 5)
Time Frame: Visit 6 (Month 5)
Population: Included all enrolled participants who were evaluable for this outcome at the specified timepoint.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 86
g/dL | 10.82 (1.64)

12. Primary Outcome: Mean Hemoglobin Value at Visit 7 (Month 6)
Time Frame: Visit 7 (Month 6)
Population: Included all enrolled participants who were evaluable for this outcome at the specified timepoint.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 78
g/dL | 10.94 (1.51)

13. Secondary Outcome: Mean Methoxy Polyethylene Glycol-Epoetin Beta Dose During the Study
Time Frame: Visit 2 (Month 1), Visit 3 (Month 2), Visit 4 (Month 3), Visit 5 (Month 4), Visit 6 (Month 5), Visit 7 (Month 6)
Population: Included all enrolled participants who were evaluable for this outcome measure and "n" represents number of participants evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 91
mcg
  Visit 2 (n=91) | 106.59 (42.79)
  Visit 3 (n=87) | 108.91 (39.80)
  Visit 4 (n=90) | 117.38 (46.53)
  Visit 5 (n=89) | 122.47 (49.72)
  Visit 6 (n=85) | 127.35 (47.50)
  Visit 7 (n=83) | 133.73 (50.67)

14. Secondary Outcome: Number of Participants With Dose Adjustments of Methoxy Polyethylene Glycol-Epoetin Beta
Description: Dose adjustment included dose increase or dose decrease with respect to previous visit's dose.
Time Frame: Visit 2 (Month 1), Visit 3 (Month 2), Visit 4 (Month 3), Visit 5 (Month 4), Visit 6 (Month 5), Visit 7 (Month 6), Visit 8 (Month 7)
Population: Included all enrolled participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 97
participants
  Visit 2-Decreased (n=97) | 0
  Visit 2-Increased (n=97) | 0
  Visit 3-Decreased (n=91) | 6
  Visit 3-Increased (n=91) | 4
  Visit 4-Decreased (n=86) | 1
  Visit 4-Increased (n=86) | 7
  Visit 5-Decreased (n=90) | 4
  Visit 5-Increased (n=90) | 18
  Visit 6-Decreased (n=88) | 3
  Visit 6-Increased (n=88) | 16
  Visit 7-Decreased (n=85) | 2
  Visit 7-Increased (n=85) | 11
  Visit 8-Decreased (n=81) | 4
  Visit 8-Increased (n=81) | 11

15. Secondary Outcome: Number of Participants Treated According to European Renal Best Practice Guideline (ERBPG) and National Kidney Function (NKF) Kidney Disease Outcomes Quality Initiative (NKF KDOQI) and Mircera Package Insert
Description: Number of participants who received treatment as per the guidelines specified by ERBPG, NKF KDOQI, and Mircera package insert were to be reported.
Time Frame: Up to 6 months
Population: Due to observational nature of the study, the data for this outcome measure could not be collected.
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: The seriousness of the adverse events was not captured in this observational study, therefore all adverse events are reported as serious adverse events.
Arm/Group | Chronic Renal Anemia Participants
Serious Adverse Events (participants affected / at risk) | 79/98
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chronic Renal Anemia Participants (N=98)
Anemia (Blood and lymphatic system disorders) | 4
Anaemia megaloblastic (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Arteriovenous fistula thrombosis (Vascular disorders) | 1
Bone marrow failure (Blood and lymphatic system disorders) | 1
Bradycardia (Cardiac disorders) | 2
Cardiac arrest (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Tachycardia (Cardiac disorders) | 1
Transient ischaemic attack (Cardiac disorders) | 1
Vascular access complication (Vascular disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Arteriovenous fistula operation (Surgical and medical procedures) | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 1
Catheter placement (Surgical and medical procedures) | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Nephrectomy (Surgical and medical procedures) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
BK virus infection (Infections and infestations) | 1
Cholecystitis acute (Infections and infestations) | 1
Colitis (Infections and infestations) | 1
Duodenitis (Infections and infestations) | 1
Gastritis (Infections and infestations) | 3
Gastroduodenitis (Infections and infestations) | 1
Helicobacter infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 4
Pyelonephritis acute (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Septic shock (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Chest pain (General disorders) | 3
Death (General disorders) | 2
Medical device complication (General disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal pain (Renal and urinary disorders) | 1
Renal mass (Renal and urinary disorders) | 1
Vitamin B1 deficiency (Metabolism and nutrition disorders) | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Depression (Psychiatric disorders) | 1
Headache (Nervous system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.